CLINICAL TRIAL: NCT01144637
Title: A Randomized, Double-Blind, Placebo-Controlled Phase III Trial to Evaluate Immunogenicity and Safety of Three Consecutive Production Lots of IMVAMUNE® (MVA-BN®) Smallpox Vaccine in Healthy, Vaccinia-Naïve Subjects
Brief Title: A Trial to Evaluate Immunogenicity and Safety of Three Consecutive Production Lots of IMVAMUNE® (MVA-BN®) Smallpox Vaccine in Healthy, Vaccinia-naïve Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: POX-MVA-013
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): Two vaccinations four weeks apart (at Day 0 and Day 28) with IMVAMUNE® Lot #1
  Interventions: Biological: IMVAMUNE®
- Group 2 (Experimental): Two vaccinations four weeks apart (at Day 0 and Day 28) with IMVAMUNE® Lot #2
  Interventions: Biological: IMVAMUNE®
- Group 3 (Experimental): Two vaccinations four weeks apart (at Day 0 and Day 28) with IMVAMUNE® Lot #3
  Interventions: Biological: IMVAMUNE®
- Group 4 (Placebo Comparator): Two vaccinations four weeks apart (at Day 0 and Day 28) with 0.5 ml Placebo, Tris-buffered saline (TBS)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IMVAMUNE® — 0.5 ml IMVAMUNE® vaccine containing at least 1 x 10E8 TCID50 (standard dose)
  Other Names: IMVANEX; MVA-BN®
  Arms: Group 1; Group 2; Group 3
Other: Placebo — 0.5 ml TBS
  Other Names: Tris-buffered-saline
  Arms: Group 4

SUMMARY:
A randomized, double-blind, placebo-controlled Phase III trial to evaluate immunogenicity and safety of three consecutive production lots of IMVAMUNE® (MVA-BN®) smallpox vaccine in healthy, vaccinia-naïve subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 18 to 40 years of age
* The subject has read, signed and dated the informed consent form, having been advised of the risks and benefits of the trial in a language understood by the subject and prior to performance of any trial specific procedures
* BMI ≥ 18.5 and < 35
* Women of childbearing potential (WOCBP) must have used an acceptable method of contraception for 30 days prior to the first vaccination, must agree to use an acceptable method of contraception during the trial, and must avoid becoming pregnant for at least 28 days after the last vaccination. A woman is considered of childbearing potential unless post-menopausal or with a history of hysterectomy (Acceptable contraception methods are restricted to abstinence, barrier contraceptives, intrauterine contraceptive devices or licensed hormonal products)
* WOCBP must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to each vaccination
* White blood cells ≥ 2,500/mm3 < ULN
* Absolute neutrophil count (ANC) within normal limits
* Hemoglobin within normal limits
* Platelets within normal limits
* Adequate renal function defined as a calculated Creatinine Clearance (CrCl) > 60 ml/min as estimated by the Cockcroft-Gault equation:

  * For men: (140 - age in years) x (body weight in kg) ÷ (serum creatinine in mg/dl x 72) = CrCl (ml/min)
  * For women: multiply the result by 0.85 = CrCl (ml/min).
* Adequate hepatic function defined as:

  * a. Total bilirubin ≤ 1.5 x ULN in the absence of other evidence of significant liver disease
  * b. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase ≤ 1.5 x ULN
* Troponin I < 2 x ULN
* Electrocardiogram (ECG) without clinically significant findings (e.g. any kind of atrioventricular or intraventricular conditions or blocks such as complete left or right bundle branch block, AV node block, QTc or PR prolongation, premature atrial contractions or other atrial arrhythmia, sustained ventricular arrhythmia, two premature ventricular contractions in a row, ST elevation consistent with ischemia)

Exclusion criteria

* Typical vaccinia scar
* Known or suspected history of smallpox vaccination
* History of vaccination with any poxvirus-based vaccine
* US Military service prior to 1991 or after January 2003
* Pregnant or breast-feeding women
* Uncontrolled serious infection, i.e. not responding to antimicrobial therapy
* History of any serious medical condition, which in the opinion of the investigator would compromise the safety of the subject or would limit the subject's ability to complete the trial
* History of or active autoimmune disease, persons with vitiligo or thyroid disease taking thyroid replacement are not excluded
* Known or suspected impairment of immunologic function including, but not limited to, HIV Infection, clinically significant liver disease (including chronic active HBV or HCV), diabetes mellitus, moderate to severe kidney impairment
* History of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure. Subjects with history of skin cancer must not be vaccinated at the previous tumor site
* History or clinical manifestation of clinically significant and severe hematological, pulmonary, central nervous, cardiovascular or gastrointestinal disorders
* Clinically significant mental disorder not adequately controlled by medical treatment
* History of coronary heart disease, myocardial infarction, angina pectoris, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, or any other heart condition under the care of a doctor
* Known history of an immediate family member (father, mother, brother, or sister) who has had onset of ischemic heart disease before age 50 years
* Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool (http://hin.nhlbi.nih.gov/atpiii/calculator.asp?usertype=prof) NOTE: This criterion applies only to subjects 20 years of age and older
* Active or history of chronic alcohol abuse and/or intravenous and/or nasal drug abuse (within the past 6 months)
* Known allergy to IMVAMUNE® vaccine and its constituents, e.g. tris (hydroxymethyl)-amino methane, including know allergy to egg or aminoglycosides
* History of anaphylaxis or severe allergic reaction to any vaccine
* Acute disease (illness with or without a fever) at the time enrollment
* Body temperature ≥100.4°F (≥38.0°C) at the time of enrollment
* Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior to or after trial vaccination
* Having received any vaccinations or planned vaccinations with a killed vaccine within 14 days prior to or after trial vaccination
* Chronic systemic administration (defined as more than 14 days) of > 5 mg prednisone (or equivalent)/day or any other immune-modifying drugs during a period starting from three months prior to administration of the vaccine and ending at last physical trial visit (V5)
* Post organ transplant subjects whether or not receiving chronic immunosuppressive therapy
* Administration or planned administration of immunoglobulins and/or any blood products during a period starting from three months prior to administration of the vaccine and ending at last physical trial visit (V5)
* Use of any investigational or non-registered drug or vaccine other than the trial vaccine within 30 days preceding the first dose of the trial vaccine, or planned administration of such a drug during the trial period
* Trial personnel

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4005 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Turner Overton, MD, Principal Investigator — Division of Infectious Diseases University of Alabama at Birmingham
Locations (34):
- United States (34):
  - Alabama Vaccine Research Clinic, Birmingham, Alabama
  - Anaheim Clinical Trials, Anaheim, California
  - National Research Institute, Los Angeles, California
  - Northern California Clinical Research Center (NCCRC), Redding, California
  - Therapeutics Clinical Research, San Diego, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Avail Clinical Research, LLC, DeLand, Florida
  - Broward Research Group, Hollywood, Florida
  - Accelovance Melbourne, Melbourne, Florida
  - Southeast Regional Research Group, Savannah, Georgia
  - Advanced Clinical Research, Inc., Meridian, Idaho
  - Accelovance Peoria, Peoria, Illinois
  - Heartland Research Associates, Augusta, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Benchmark Research, Metairie, Louisiana
  - QPS Bio-Kinetic, Springfield, Missouri
  - Washington University in St. Louis, School of Medicine, St Louis, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Clinical Research Center of Nevada, LLC, Las Vegas, Nevada
  - Rochester Clinical Research, Inc., Rochester, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Family Practice Center of Wooster, Wooster, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Columbia Research Group, Inc., Portland, Oregon
  - Omega Medical Research, Warwick, Rhode Island
  - PMG Research of Charleston, Mt. Pleasant, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Benchmark Research, Fort Worth, Texas
  - Tanner Clinic, Layton, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - University Physicians Internal Medicine University Physicians & Surgeons, Inc., Huntington, West Virginia

REFERENCES:
- [Derived] Overton ET, Lawrence SJ, Wagner E, Nopora K, Rosch S, Young P, Schmidt D, Kreusel C, De Carli S, Meyer TP, Weidenthaler H, Samy N, Chaplin P. Immunogenicity and safety of three consecutive production lots of the non replicating smallpox vaccine MVA: A randomised, double blind, placebo controlled phase III trial. PLoS One. 2018 Apr 13;13(4):e0195897. doi: 10.1371/journal.pone.0195897. eCollection 2018. PMID 29652929

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 999 | 1005 | 999 | 1002
Completed (active trial phase) | 925 | 929 | 939 | 946
Not Completed | 74 | 76 | 60 | 56

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 999 | 1005 | 999 | 1002 | 4005
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (6.28) | 27.5 (6.24) | 28.0 (6.31) | 27.7 (6.38) | 27.7 (6.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 526 | 527 | 494 | 539 | 2086
  Male | 473 | 478 | 505 | 463 | 1919

OUTCOME MEASURES:

1. Primary Outcome: PRNT GMT
Description: Geometric Mean Titers (GMT) based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Titers below the detection limit are included with a value of '1'.
Time Frame: 2 weeks following the second vaccination
Population: Per-protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 637 | 628 | 641 | 643
Titer | 110.7 [103.4 to 118.4] | 100.5 [93.7 to 107.8] | 117.2 [109.0 to 126.0] | 1.0 [1.0 to 1.1]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Equivalence — The equivalence margins to show that the 3 vaccine lots are equivalent in terms of PRNT GMTs at Week 6 was predefined as [0.5; 2] for the GMT ratios (pairwise); GMT ratio (Group 1 / Group 2) = 1.1012, 95% CI 2-sided [0.9992 to 1.2136]
Statistical Analysis 2: Comparison: Group 1 vs Group 3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (Group 1 / Group 3) = 0.9444, 95% CI 2-sided [0.8554 to 1.0427]
Statistical Analysis 3: Comparison: Group 2 vs Group 3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT ratio (Group 2 / Group 3) = 0.8577, 95% CI 2-sided [0.7753 to 0.9488]

2. Secondary Outcome: ELISA GMT
Description: Geometric Mean Titers (GMT) based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Titers below the detection limit are included with a value of '1'.
Time Frame: 2 weeks following the second vaccination
Population: Per-protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 637 | 628 | 641 | 643
Titer | 901.0 [844.8 to 961.1] | 794.4 [738.1 to 855.0] | 946.7 [888.2 to 1008.9] | 1.2 [1.1 to 1.3]

3. Secondary Outcome: PRNT Seroconversion Rate
Description: Seroconversion rate based on Plaque Reduction Neutralization Test (PRNT). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (2) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: 2 weeks following the second vaccination
Population: Per-protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 637 | 628 | 641 | 643
percentage of subjects | 99.8 [99.1 to 100.0] | 99.7 [98.9 to 100.0] | 99.8 [99.1 to 100.0] | 1.4 [0.6 to 2.6]

4. Secondary Outcome: ELISA Seroconversion Rate
Description: Seroconversion rate based on Enzyme-linked Immunosorbent Assay (ELISA). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (50) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: 2 weeks following the second vaccination
Population: Per-protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 637 | 628 | 641 | 643
percentage of subjects | 99.7 [98.9 to 100.0] | 99.5 [98.6 to 99.9] | 100.0 [99.4 to 100.0] | 2.0 [1.1 to 3.4]

5. Secondary Outcome: Correlation PRNT vs ELISA Titers
Description: Pearson Correlation Coefficient between the log10 transformed PRNT titers and the log10 transformed ELISA titers
Time Frame: 2 weeks following the second vaccination
Population: Per-protocol Set
Measure: Number (95% Confidence Interval); unit: Pearson correlation coefficient
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 637 | 628 | 641 | 643
Pearson correlation coefficient | 0.581 [0.527 to 0.630] | 0.620 [0.569 to 0.666] | 0.612 [0.561 to 0.658] | 0.486 [0.424 to 0.543]

6. Secondary Outcome: Serious Adverse Events
Description: Incidence, relationship and intensity of any Serious Adverse Event (SAE)
Time Frame: within 30 weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 999 | 1005 | 999 | 1002
Participants
  Any SAE | 11 | 7 | 7 | 8
  Any SAE with intensity >= Grade 3 | 8 | 6 | 6 | 5
  Any SAE assessed as related to vaccine | 0 | 0 | 0 | 1

7. Secondary Outcome: Cardiac Signs or Symptoms
Description: Incidence, relationship and intensity of any cardiac sign or symptom indicating a case of myo-/pericarditis (Adverse Event of Special Interest (AESI)).
  An AESI was defined in this trial as:
  * Any cardiac sign or symptom developed since the first vaccination
  * ECG changes determined to be clinically significant
  * Cardiac enzyme Troponin I >= 2 x ULN (>= Grade 2)
Time Frame: within 30 weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 999 | 1005 | 999 | 1002
Participants
  Any AESI | 2 | 5 | 1 | 1
  Any AESI with intensity >= Grade 3 | 0 | 0 | 0 | 0
  Any AESI assessed as related to vaccine | 0 | 1 | 1 | 0

8. Secondary Outcome: Related Grade >=3 Adverse Events
Description: Incidence of any Grade >=3 Adverse Events probably, possibly or definitely related to the trial vaccine. Pooled solicited (general only) and unsolicited AEs
Time Frame: within 29 days after any vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 999 | 1005 | 999 | 1002
Participants | 58 | 57 | 53 | 27

9. Secondary Outcome: Unsolicited Non-serious AEs: Intensity
Description: Occurrence of unsolicited non-serious AEs by Intensity
Time Frame: within 29 days after any vaccination
Population: Full Analysis Set
Measure: Number; unit: events
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 999 | 1005 | 999 | 1002
events
  Total | 288 | 350 | 320 | 280
  Grade 1 | 190 | 236 | 218 | 192
  Grade 2 | 88 | 100 | 94 | 82
  Grade 3 | 10 | 14 | 8 | 6
  Grade 4 | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 0 | 0

10. Secondary Outcome: Unsolicited Non-serious AEs: Relationship to Vaccination
Description: Occurrence of unsolicited non-serious AEs by relationship to study vaccine
Time Frame: within 29 days after any vaccination
Population: Full Analysis Set
Measure: Number; unit: events
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 999 | 1005 | 999 | 1002
events
  Unrelated/None | 187 | 218 | 181 | 189
  Unlikely | 40 | 56 | 61 | 51
  Possible | 28 | 42 | 34 | 29
  Probable | 5 | 6 | 7 | 6
  Definite | 28 | 27 | 35 | 4
  Missing | 0 | 1 | 2 | 1
  Total | 288 | 350 | 320 | 280

11. Secondary Outcome: Solicited Local AEs
Description: Incidence and intensity of solicited local AEs (redness, swelling, induration, pruritus and pain). Percentages based on subjects with at least one completed diary card.
Time Frame: within 8 days after any vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 985 | 976 | 982 | 980
Participants
  Pain: Any | 846 | 823 | 830 | 187
  Pain: Grade >=3 | 76 | 66 | 76 | 10
  Erythema: Any | 597 | 610 | 581 | 173
  Erythema: Grade >=3 | 15 | 18 | 12 | 0
  Swelling: Any | 508 | 513 | 499 | 55
  Swelling: Grade >=3 | 9 | 10 | 4 | 0
  Induration: Any | 454 | 439 | 442 | 45
  Induration: Grade >=3 | 4 | 4 | 2 | 0
  Pruritis: Any | 430 | 424 | 414 | 115
  Pruritis: Grade >=3 | 20 | 15 | 13 | 2

12. Secondary Outcome: Solicited General AEs
Description: Incidence of solicited general AEs (pyrexia, headache, myalgia, chills, nausea, and fatigue): Intensity and relationship to vaccination. Percentages based on subjects with at least one completed diary card.
Time Frame: within 8 days after any vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 985 | 976 | 982 | 980
Participants
  Pyrexia: Any | 17 | 19 | 14 | 9
  Pyrexia: Related | 13 | 15 | 14 | 6
  Pyrexia: Grade >=3 | 2 | 4 | 1 | 0
  Headache: Any | 321 | 349 | 354 | 251
  Headache: Related | 279 | 314 | 318 | 208
  Headache: Grade >=3 | 28 | 24 | 20 | 21
  Myalgia: Any | 425 | 403 | 431 | 172
  Myalgia: Related | 404 | 381 | 414 | 156
  Myalgia: Grade >=3 | 25 | 25 | 27 | 7
  Chills: Any | 108 | 108 | 90 | 57
  Chills: Related | 96 | 96 | 84 | 51
  Chills: Grade >=3 | 10 | 7 | 12 | 3
  Nausea: Any | 166 | 179 | 163 | 128
  Nausea: Related | 146 | 158 | 144 | 99
  Nausea: Grade >=3 | 13 | 16 | 16 | 12
  Fatigue: Any | 305 | 303 | 287 | 201
  Fatigue: Related | 276 | 279 | 267 | 176
  Fatigue: Grade >=3 | 32 | 27 | 29 | 13

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
All-Cause Mortality (participants affected / at risk) | 1/999 | 0/1005 | 0/999 | 0/1002
Serious Adverse Events (participants affected / at risk) | 11/999 | 7/1005 | 7/999 | 8/1002
Other Adverse Events (participants affected / at risk) | 53/999 | 70/1005 | 65/999 | 48/1002
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=999) | Group 2 (N=1005) | Group 3 (N=999) | Group 4 (N=1002)
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 2
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=999) | Group 2 (N=1005) | Group 3 (N=999) | Group 4 (N=1002)
Injection site haematoma (General disorders) | 5 | 11 | 8 | 5
Injection site induration (General disorders) | 14 | 15 | 21 | 0
Nasopharyngitis (Infections and infestations) | 11 | 14 | 11 | 3
Upper respiratory tract infection (Infections and infestations) | 17 | 21 | 20 | 31
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 6 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes